CLINICAL TRIAL: NCT06743373
Title: Cannabis Effects on Sleep, Circadian Rhythms, and Light Sensitivity in Young Adults (CASCILS)
Brief Title: Cannabis Effects on Sleep, Circadian Rhythms, and Light Sensitivity in Young Adults
Acronym: CASCILS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Brant Hasler, Associate Professor of Psychiatry, Psychology, and Clinical and Translational Science, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY24050074; 1R01DA061223-01 (NIH)
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cannabis Use; Sleep; Circadian Rhythm
Keywords: cannabis; sleep; circadian rhythms; photosensitivity; cannabis discontinuation
MeSH Terms: conditions — Marijuana Abuse; Photosensitivity Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabis-Using (Experimental): The cannabis-using arm will consist of 60 young people reporting regular cannabis use. Participants will complete a 1-week baseline protocol followed by a 4-week cannabis discontinuation protocol (intervention).
  Interventions: Behavioral: Cannabis Discontinuation
- Control (No Intervention): The control arm will consist of 30 young people without current cannabis use. Participants will complete a 1-week baseline protocol. No intervention will be administered.

INTERVENTIONS:
Behavioral: Cannabis Discontinuation — Cannabis-using participants will participate in an orientation session with a clinician and asked to abstain from cannabis use for four weeks, using established procedures for abstinence monitoring and reinforcement.
  Arms: Cannabis-Using

SUMMARY:
The goal of this study is to learn how cannabis use and discontinuation affect sleep, circadian rhythms, and sensitivity to light. The main questions it aims to answer are:

1. Does cannabis use and discontinuation impact sleep drive?
2. Does cannabis use and discontinuation impact light sensitivity and circadian phase?

DETAILED DESCRIPTION:
Researchers will compare sleep, circadian phase, and light sensitivity within regular cannabis users before, during, and after a cannabis discontinuation protocol; researchers will also compare sleep, circadian phase, and light sensitivity between regular cannabis users and control non-cannabis users.

Participants will:

1. Participate in a 1-week baseline period consisting of at-home monitoring (sleep diaries, actigraphy, EEG headband).
2. Participate in a 2-night lab visit consisting of circadian phase and light sensitivity assessment.
3. Participate in a 4-week cannabis discontinuation protocol (cannabis users only).
4. Participate in a second 2-night lab visit after the discontinuation protocol (cannabis users only).

ELIGIBILITY:
List the inclusion criteria:

* Age 18-25 years
* Physically and psychiatrically healthy, as determined by instruments described below
* Cannabis-Using group only: Regular cannabis use, defined as "frequent" (6-29 days/month) or "daily" (daily) use over the past 3 months
* Cannabis-Using group only: Willingness to discontinue cannabis for 4 weeks.
* Control group only: No cannabis use in the past 3 months. Deny engaging in daily or near-daily cannabis use during the past year. No history of alcohol and/or substance use disorders. No current sleep disorders (including insomnia and delayed sleep phase disorder).
* Provision of written informed consent

List the exclusion criteria:

* Significant or unstable acute or chronic medical conditions. Examples of such conditions include, but are not limited to, central nervous system disorders (e.g., head injury, seizure disorder, multiple sclerosis, tumor), cardiovascular or hemodynamically significant cardiac disease, liver disease (e.g., acute or chronic hepatitis, hepatic insufficiency), migraine or chronic headaches, active peptic ulcer disease, inflammatory bowel disease, renal failure, arthritis, and diabetes and other endocrine disorders. Seizure disorder in particular will be exclusionary due to the increased risk it confers for cannabis withdrawal symptoms. Eye/retinal conditions such as diabetic retinopathy or glaucoma will be exclusionary, although should be very rare in this population. Individuals with well-controlled health conditions that do not affect sleep, retinal function, and/or well-being (e.g., well-controlled thyroid disorders, asthma, or ulcer) will not be excluded. To evaluate these criteria, potential participants will complete a locally-developed Medical History Questionnaire.
* Past or current DSM-5 bipolar disorder or psychotic disorders. Psychiatric disorders will be evaluated using the Mini International Neuropsychiatric Interview (MINI) and the WHO-DAS 2.0, supplemented by clinical interview. We will not exclude participants for subsyndromal symptoms or disorders in these domains. We will not exclude participants for other psychiatric disorders, particularly given the high comorbidity between cannabis use disorder and major depression and anxiety disorder, as long as severity is in the moderate range or lower based on the WHO-DAS 2.0 (average score <4).
* Daily use of alcohol; regular use of illicit substances. Regular use (as defined above) of illicit substances other than cannabis over the past 3 months will be exclusionary. Substance use will be assessed using the Timeline Follow Back method, as well as a urine drug screen.
* Past or current substance use disorders other than cannabis use disorder, nicotine use disorder, and mild alcohol use disorder (moderate and severe alcohol use disorder are exclusionary).
* Current syndromal sleep disorders other than insomnia and delayed sleep phase disorder, including narcolepsy, restless legs syndrome, obstructive sleep apnea, and current night shift work (i.e., any work occurring between the hours of midnight and 6:00 a.m.). We will not exclude for subsyndromal symptoms or disorders in these domains. We will not exclude Cannabis-using participants for insomnia and delayed sleep phase disorder because of their conceptual overlap and high co-occurrence with sleep phenotypes of interest. Sleep disorders will be diagnosed according to criteria in the DSM-5 and the International Classification of Sleep Disorders, 3rd Edition, 2014. These disorders will be evaluated using clinical interview and the locally-developed Structured Clinical Interview for Sleep Disorders. Control participants will be excluded for any current sleep disorders, including insomnia and delayed sleep phase disorder.
* Travel across 2+ time zones in the past 60 days.
* Benzodiazepines and non-benzodiazepine hypnotic drugs ("Z-drugs"). Other sleep-promoting medications will be permitted, including SSRIs/SNRIs, will be permitted if on stable dose and not in the acute phase of treatment. In order to evaluate medications, participants will complete a listing of current medications, including prescription and over the counter medications, "natural" preparations, and nutritional supplements.
* Individuals with a Pennsylvania Medical Marijuana Card using dispensary-obtained marijuana or other THC products for documented Qualifying Medical Conditions other than those of a mental health nature will be excluded. However, individuals who have been issued a Pennsylvania Medical Marijuana ID card for a mental health condition will not be excluded from the study.

There will not be any Medical Record review. For most individuals, the Medical History Questionnaire, including medical conditions and medications, will be sufficient for identifying exclusionary medical criteria. For instances where an individual is uncertain about exclusionary or current medical conditions or medications, medical records, prescription records or labeled prescription pill bottles, or a Release of Information to contact the individual's Primary Care Practitioner [PCP] to clarify the individual's medical status will be obtained.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Homeostatic Sleep Drive | Baseline, 1 week
  Rate of slow wave activity dissipation, assessed by at-home EEG headband. Compared within person (cannabis-using days vs. non using days), between groups (Cannabis-Using, Control) at Baseline, and within-group (Cannabis-Using) between Baseline and Post-discontinuation.
Circadian Photosensitivity | Discontinuation, 4 weeks
  Light-Induced Melatonin Suppression. Melatonin levels on during a 60-minute light exposure will be compared to melatonin levels on a prior night under dim light conditions (when the dim light melatonin onset was assessed). The primary outcome will be % reduction in melatonin levels. Will be compared between groups (Cannabis-Using, Control) at Baseline and within-group (Cannabis-Using) between Baseline and Post-discontinuation.
Retinal Responsivity | End of discontinuation, 4 weeks
  Retinal responsivity assessed via pupillometry (specifically the Post-Illumination Pupil Response; PIPR). Will be compared between groups (Cannabis-Using, Control) at Baseline and within group (Cannabis-Using.

SECONDARY OUTCOMES:
Circadian phase | End of discontinuation, 4 weeks
  Dim light melatonin onset (DLMO). Compared between groups (Cannabis-Using, Control) at Baseline, and within-group (Cannabis-Using) between Baseline and Post-discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Brant P Hasler, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Hospital (Thomas Detre Hall), Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers are currently requesting permission from NIDA to share de-identified data via the National Sleep Research Resource (NSRR), which will determine in part which IPD are included. Researchers anticipate sharing, at a minimum, participant's sociodemographic characteristics and the data required to test our listed primary and secondary aims, including substance use data, as well as data from wrist actigraphy, sleep electroencephalography (EEG), salivary melatonin data, and pupillometry.
Supporting Information: Study Protocol
Time Frame: If researchers use the NSRR as planned, the research community will have access to data at the end of the grant award and/or when a publication has been submitted. Once the data are submitted to NSRR, the NSRR platform will control the long-term persistence of the data set. Currently, NSRR has no process for deleting or retiring data sets and has created a stable and sustainable infrastructure that will allow currently hosted data to stay available through the lifetime of the repository.
Access Criteria: To request access to study data on the NSRR, researchers would use the standard processes that includes research proposal submission and review by the NSRR Data Access Review Committee. The standard NSRR data access process allows time limited access and is renewable. Written requests from qualified investigators will be submitted on a standardized data request and analysis form, which will then be reviewed by PI Hasler. All data requests will be logged in a repository tracking log. IRB and/or Data Use Agreements (as appropriate) will be put in place before any transfer of data. Investigators receiving the data much abide by the conditions of these agreements.